CLINICAL TRIAL: NCT02066259
Title: OctavaColon Blood Tests OctavaGold and OctavaSilver - Blood Tests for the Help in Diagnosis of Colon Cancer Clinical Study Protocol
Brief Title: OctavaColon Cancer Blood Tests OctavaGold and OctavaSilver - Blood Tests for the Help in Diagnosis of Colon Cancer Clinical Study Protocol
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Eventus Diagnostics Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: OctavaColon_001
Record Dates: First submitted 2014-02-09; First posted 2014-02-19 (Estimated); Last update posted 2014-08-05 (Estimated); Status verified 2014-08

CONDITIONS: Colon Cancer
Keywords: colon cancer; cancer associated auto antibodies; colon cancer blood test
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Human plasma samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- healthy_0: healthy, people with normal (negative) colonoscopy results.
- patient_1: people with biopsy/surgery verified carcinoma of the colon, either an Adenocarcinoma, or carcinoma in situ
- benign_2: people with biopsy verified benign polyps of the colon one of the following - Villus adenoma, Tubular adenoma, Low grade dysplasia, Intermediate grade dysplasia, High grade dysplasia, Severe dysplasia

SUMMARY:
The OctavaColon tests are qualitative plasma tests that are indicated to people above 18 years of age suspected with colon abnormality. The blood tests will provide additional information to the doctor in the course of colon cancer diagnosis for both normal population and high risk population

DETAILED DESCRIPTION:
The clinical objective of this study is to develop two antibody-based blood tests for additional information during colon cancer diagnosis -

1. Highly specific (OctavaGold) - provides additional information to doctors during evaluation of normal population.
2. Highly sensitive (OctavaSilver) - provides additional information to doctors during evaluation of high risk population.

The study will be considered successful it can achieve at least one of the following sets of performances -

1. For the OctavaGold - 95% specificity with at least 50% sensitivity.
2. For the OctavaSilver - 95% sensitivity with at least 50% specificity. The biological objective of this study is to find the best set of antigens, that when combined with the appropriate algorithm will support each of the above clinical objectives

ELIGIBILITY:
Inclusion Criteria:

Subjects 18 years or over. Subjects scheduled for colonoscopy or surgery

Exclusion Criteria:

* Subjects less than 18 years of age
* Previous or concurrent synchronous cancers other than previous malignancies of the colon and recovered melanoma
* Autoimmune disorders diagnosed subjects
* Hematological malignancies
* Subjects under active chemotherapy treatment or chemotherapy in the past 6 months
* Steroid treatment in the past 3 months
* Subject undergoing immunosuppressive treatments
* Subject with verified melanoma colon cancer
* Subject with verified sarcoma colon cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: There are 3 different populations that will participate in the study-
  1. Any person with suspected colon abnormality, that will be classified after colonoscopy/surgery as "colon cancer patient" will be a part of group1 - "Patient".
  2. Any person with suspected colon abnormality, that will be classified after colonoscopy as "benign polyp" will be a part of group2 - "benign".
  3. Any person with suspected colon abnormality, that will be classified after colonoscopy as "normal/healthy" will be a part of group0 - "healthy".
Sampling Method: Probability Sample
Enrollment: 1080 (Estimated)
Dates: Start 2014-08; Primary Completion 2016-03 (Estimated); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
Number of participants in each of the clinicaly defined groups (0,1 and 2). | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Galit Yahalom, Ph.D., Study Director — Eventus Dx
Locations (3):
- Israel (3):
  - Soroka Medical Center, Beersheba
  - "Carmel" Medical Center, Haifa
  - Sheba Tel hashomer, Ramat Gan

REFERENCES:
- [Background] Yahalom G, Weiss D, Novikov I, Bevers TB, Radvanyi LG, Liu M, Piura B, Iacobelli S, Sandri MT, Cassano E, Allweis TM, Bitterman A, Engelman P, Vence LM, Rosenberg MM. An Antibody-based Blood Test Utilizing a Panel of Biomarkers as a New Method for Improved Breast Cancer Diagnosis. Biomark Cancer. 2013 Nov 19;5:71-80. doi: 10.4137/BIC.S13236. eCollection 2013. PMID 24324350